CLINICAL TRIAL: NCT03469713
Title: Nivolumab Plus Stereotactic Body Radiotherapy (SBRT) in II and III Line of Patients With Metastatic Renal Cell Carcinoma (mRCC)
Brief Title: Nivolumab Plus Stereotactic Body Radiotherapy in II and III Line of Patients With Metastatic Renal Cell Carcinoma
Acronym: NIVES
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Oncologico Italiano di Ricerca Clinica (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOIRC-06-2016
Record Dates: First submitted 2018-02-08; First posted 2018-03-19 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2021-12

CONDITIONS: Renal Cancer Metastatic
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nivolumab (Experimental): Hypofractionated radiation will be administered to a metastatic disease site at a dose and schedule of 30 Gy in 3 consecutive fractions. The day of first administration of Nivolumab will be designated as Time 1. Nivolumab will be given as flat dose of 240 mg in intravenous infusion beginning on day 1 every 14 days for 6 months, than switch to 480 mg q4-weekly in responding (CR, PR, SD) patients until PD or unacceptable toxicity .
  SRT will be administered between the first and second administration of Nivolumab (7 days after the first infusion of Nivolumab).
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Hypofractionated radiation will be administered to a metastatic disease site at a dose and schedule of 30 Gy in 3 consecutive fractions. The day of first administration of Nivolumab will be designated as Time 1. Nivolumab will be given as flat dose of 240 mg in intravenous infusion beginning on day 1 every 14 days for 6 months, than switch to 480 mg q4-weekly in responding (CR, PR, SD) patients until PD or unacceptable toxicity .
  SRT will be administered between the first and second administration of Nivolumab (7 days after the first infusion of Nivolumab).

SUMMARY:
NIVES study is an ongoing phase II, single arm, multicenter study. In this trial pts received SBRT to one non-brain measurable lesion and concomitant NIVOLUMAB, an anti-programmed cell death (PD-1). Combining SBRT with NIVO may enhance the antitumor immune responses and improve clinical outcomes, how it was demonstrated for other solid tumors with a phenomenon known as the abscopal effect . It was planned to enrolled a total of 68 pts within 12 months. The objective of the current analysis is to describe the first report of safety profile of NIVO in combination with SBRT.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years on day of signing informed consent
* Performance status of 0, 1 on the ECOG Performance Scale
* Histologically confirmed metastatic RCC not suitable for curative-intent local therapy
* Disease progressed after ≤ 2 prior anti-angiogenic therapies
* Life expectancy > 12 weeks
* 2 or more measurable non-brain sites of disease based on RECIST 1.1, whose at least one potentially suitable for treatment with SBRT. In the case of a non measurable bone lesion suitable for treatment with SBRT, even only one measurable non-brain site of disease is allowed
* Patients are eligible if CNS metastases are treated and patients have neurologically returned to baseline (except for residual signs or symptoms related to the CNS treatment) for at least 14 days prior to enrollment. In addition, patients must either be off corticosteroids or on a stable dose or decreasing dose of ≤ 10 mg daily prednisone (or equivalent)
* Adequate organ function

Exclusion Criteria:

* Prior therapy with an agent directed at PD-1, PD-L1, or PD-L2
* Currently participating in or has participated in a study of an investigational agent or using an investigational device within 2 weeks of the first dose of treatment
* Any active or recent history of a known or suspected autoimmune disease or recent history of a syndrome that required systemic corticosteroids (> 10 mg daily prednisone equivalent) or immunosuppressive medications except for syndromes which would not be expected to recur in the absence of an external trigger
* Any condition requiring systemic treatment with corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days prior to first dose of study drug. Inhaled steroids and adrenal replacement steroid doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease
* Active brain (CNS) metastases and/or carcinomatous meningitis
* Prior monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent. Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 14 days prior to the first dose of trial treatment
* Any positive test for hepatitis B or hepatitis C virus indicating acute or chronic infection
* Additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy
* Evidence of interstitial lung disease, active non-infectious pneumonitis, or a history of grade 3 or greater pneumonitis
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness
* Live vaccine within 30 days prior to the first dose of trial treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2019-03-04 (Actual); Study Completion 2021-07-14 (Actual)

PRIMARY OUTCOMES:
ORR Objective Response Rate | 36 months from the first administration of nivolumab
  Objective Response Rate (ORR) , as determined by investigator assessment per RECIST 1.1 Secondary as determined by investigator assessment per RECIST 1.1

SECONDARY OUTCOMES:
PFS Progression Free Survival | 36 months from the first administration of nivolumab
  the time between the date of registration and the first date of documented progression, based on invesigator assessment (as per RECIST 1.1 criteria), or death due to any cause, whichever occurs first
OS Overall Survival | 36 months from the first administration of nivolumab
  the time from registration to the date of death from any cause
ORR (Objective Response Rate) of irradiated and non-irradiated metastases and duration of response | 36 months from the first administration of nivolumab
  determined by investigator assessment per RECIST 1.1
Incidence, nature and severity of Adverse Event (safety and tolerability) | 36 months from the first administration of nivolumab
  All Adverse Events (AEs) and laboratory abnormalities will be collected and graded by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v. 4.03

OTHER OUTCOMES:
Analysis of expression of PD-L1 | 36 months from the first administration of nivolumab
  Immune checkpoint inhibitors act by shortcutting the communication between immune cells and tumor cells mediated by the PD1-PDL1 interaction. Discordant results about the correlation of PDL1 expression and response to immunotherapy exist. Thus, we will investigate the expression of PDL1 in the tumor using four available IHC test (Dako 28.8, Dako 22C3, Ventana SP142, Ventana SP 263) and we will correlate levels of expression with response to treatment.
Analysis of the genetic background of the tumor and its impact on the response to therapy | 36 months from the first administration of nivolumab
  To evaluate whether and how the initial genetic background of the renal carcinoma may impact on response to treatment in the present setting a deep sequencing analysis will be performed to assess mutational status of 578 cancer genes using the Comprehensive Cancer Design panel (Roche) and MySeq Illumina Next Generation Sequencer. The overall mutations load and the type of mutations detected will be correlated with the response to treatment.
Analysis of the immuno-modulation during therapy. | 36 months from the first administration of nivolumab
  To investigate the effect of stereotactic radiotherapy on the modulation of the immune system we propose to analyze variation in the plasma levels of soluble immune-modulators during treatment. Will be use the Bio-Plex Pro™ Human Inflammation Assay (Bioplex, Biorad) that enables to detect and quantify a panel of 24 key biomarkers of inflammation including TNF superfamily proteins, IFN family proteins, and Treg cytokines
Identification of somatic mutations associated with acquired resistance to checkpoint inhibitors | 36 months from the first administration of nivolumab
  we will investigate JAK1, JAK2 and B2M mutations by in the circulating free tumor DNA (ctDNA) obtained from the plasma samples. The ctDNA will be analyzed with a multiplexed sequencing assay that generates reads containing targeted regions along with a molecular tag that allows the accompanying optimized variant analysis software to assemble the reads into families of molecules originating from the same initial ctDNA molecules and model errors accumulated during library amplification, templating, and sequencing to accurately reconstruct the sequence of the original ctDNA molecule. The resulting sequence is then used to make variant calls down to 0.05% allele ratio with high sensitivity and specificity.

CONTACTS AND LOCATIONS:
Overall Officials: Carmine Pinto, MD, Principal Investigator — Gruppo Oncologico Italiano di Ricerca Clinica
Locations (1):
- Struttura Complessa di OncologiaIRCCS- Istituto in Tecnologie Avanzate e Modelli Assistenziali in Oncologia Arcispedale Santa Maria Nuova, Reggio Emilia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maia MC, Salgia M, Pal SK. Harnessing cell-free DNA: plasma circulating tumour DNA for liquid biopsy in genitourinary cancers. Nat Rev Urol. 2020 May;17(5):271-291. doi: 10.1038/s41585-020-0297-9. Epub 2020 Mar 17. PMID 32203306